CLINICAL TRIAL: NCT04495530
Title: What Information do Patients and Carers Need to Make an Informed Decision to Commence and Discontinue Parenteral Nutrition, in Advanced Cancer?
Brief Title: Information Needs Around Parenteral nUTrition in Cancer
Acronym: INPUT
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: St George's University Hospitals NHS Foundation Trust (Other); University College London Hospitals (Other); University of Southampton (Other); London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 5217
Record Dates: First submitted 2020-07-21; First posted 2020-08-03 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Cancer; End Stage Cancer; Terminal Cancer; Neoplasms; Tumor; Malignancy; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Patients will be considering commencing or discontinuing parenteral nutrition, or will be receiving home parenteral nutrition
  Interventions: Other: Non-interventional study
- Carer: Carers will be those caring for a patient with advanced cancer who is considering commencing or discontinuing parenteral nutrition, or already receiving parenteral nutrition. Carers will also be recruited if they previously cared for a person with advanced cancer receiving parenteral nutrition in the last 12 months
  Interventions: Other: Non-interventional study

INTERVENTIONS:
Other: Non-interventional study — semi-structured interviews will take place on one occasion with participants in this study. This is qualitative research, and does not involve any interventions

SUMMARY:
This study will explore the information needs of patient's with advanced cancer, and their carers, when making a decision to commence or discontinue parenteral nutrition. Interviews will be conducted with both patients with advanced cancer, and their carers to determine the information they need to make a shared decision with the healthcare team.

DETAILED DESCRIPTION:
Parenteral nutrition (PN) is a type of nutritional liquid that is given directly into a vein, and is usually given when a person does not have a working gut. This type of nutrition is managed by a team of healthcare professionals and requires regular monitoring, such as bloods tests, to allow the team to provide the right balance of nutrients to the individual patient. This is an important decision, and the benefits, risks and consequences of having this type of nutrition should be fully explained to the patient and carer, to make sure they can make an informed decision. The aim of this study is to find out what information both patients and carers feel they need to be able to make a decision to start, and a later date stop, parenteral nutrition, with a diagnosis of advanced (incurable) cancer.

It is not clear if patients and carers get all the information they need before making this decision, and often the decision is made by a doctor and other healthcare professionals. However, patients and carers have a right to make decisions about their care. We will therefore interview patients and carers who have experience of making this decision, or in the process of making this decision, to find out what information is important to them. Our aim is to use the results from this research to improve the experience that patients and carers have in the future.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and over
* Fluent English speaker
* Is aware of diagnosis of advanced cancer
* Patient considering starting PN, is currently receiving PN or has previously received PN OR
* Carer of a patient considering, receiving or who has received PN
* NHS patient
* Assessed as having capacity to give consent and participate
* Current patient at one of the recruiting hospital sites

Exclusion Criteria:

* Private patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the inpatient and outpatient setting (intestinal failure clinic). Carers may be recruited from participating hospitals if they are caring for a patient under the care of that centre. Carers will also be recruited via social media, and online support networks.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The type of information that patients and carers need to make an informed decision to commence or discontinue parenteral nutrition | Through completion of study; expected 1 year
  This exploratory study will provide insight into the information that patients with advanced cancer, and their carers need to make an informed decision to commence and discontinue parenteral nutrition

SECONDARY OUTCOMES:
How healthcare professionals should deliver information to patients and carers in order for them to make an informed decision to commence or discontinue parenteral nutrition | Through completion of study; expected 1 year
  Patients and carers will provide insight into how they would like to receive information regarding parenteral nutrition from the clinical team. This may be through verbal or written communication.

CONTACTS AND LOCATIONS:
Overall Officials: Clare Shaw, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - St Mark's Hospital, London
  - University College London Hospitals NHS Foundation Trust, London
  - St George's NHS Foundation Trust, London
  - Royal Marsden Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No